CLINICAL TRIAL: NCT02021357
Title: The Influence of Proprioceptive Treatment for the Intensity of Pain, Muscle Activity, Level of Severity and Mandible Mobility in Individuals With Temporomandibular Dysfunction: Clinical Trial, Randomized, Controlled, Double-Blind
Brief Title: Proprioceptive Treatment for Temporomandibular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Doctor of Anatomy, University of Nove de Julho
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-2205-AR
Record Dates: First submitted 2013-12-19; First posted 2013-12-27 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Facial Pain
Keywords: Facial Pain; Physical Therapy Modalities; Temporomandibular Joint Disorders; Exercise Therapy
MeSH Terms: conditions — Facial Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hyperbolid combined with tongue exercises on the palate (Experimental): The proprioceptive treatment protocol if run in the use of exercises with hyperboloid based on studies of Biasotto-Gonzalez (2005), for each exercise will be held 6 sets of 6 reps. Between exercises, 1 minute will be established for rest of the volunteer, in order to avoid muscle fatigue and possible exacerbation of pain, and after that period you will be asked to volunteer the proprioceptive exercise of ´ ´ tongue on the hard palate ´ ´ Biasotto-Gonzalez-based (2005), which consists of the language supported in the hard palate, you must open and close the mouth, having as the principle language as a physical reference.
  Interventions: Behavioral: hyperbolid combined with tongue exercises on the palate
- Hyperbolid (Active Comparator): The proprioceptive treatment protocol if run in the use of the hyperboloid, based on studies of Biasotto-Gonzalez (2005), but without the proprioceptive exercise of language in ´ ´ hard palate ´ ´.
  For each exercise will be held 6 series of 6 repetitions, and between exercises, 1 minute will be established for rest of the volunteer, in order to avoid muscle fatigue and possible exacerbation of pain.
  Interventions: Other: hyperbolid
- Control (No Intervention): The individuals in control group did not receive any type of intervention, being offered proprioceptive treatment after the study period.

INTERVENTIONS:
Behavioral: hyperbolid combined with tongue exercises on the palate
  Arms: Hyperbolid combined with tongue exercises on the palate
Other: hyperbolid
  Arms: Hyperbolid

SUMMARY:
The project aims to assess the effects of proprioceptive treatment through the use of hyperbolid mastication apparatus on pain intensity, muscle activity and joint mobility in subjects with TMD. A randomized, blind, clinical trial will be conducted. Volunteers aged between 18 and 40 years will be recruited, with a diagnosis of muscle- and joint-related TMD according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC / TMD), being randomly divided in three different groups: Group 1 (G1) - treated with HB device combined with tongue exercises on the palate; Group 2 (G2) - treated HB alone and Group 3 (G3) - control. Treatment protocols will be applied for 12 sessions, the volunteers will be evaluated in two stages: before applying the treatment and after the last session.

DETAILED DESCRIPTION:
The temporomandibular disorder (TMD) are characterized by a set of clinical abnormalities involving the masticatory muscles, the temporomandibular joint (TMJ) and other associated structures. Several studies have supported the use of physical therapy in the treatment of this condition, especially electrotherapy, laser therapy and manual resources. However, despite advances in the search for scientific evidence, it is necessary to prove to other commonly used clinical measures in subjects with TMD, such as the use of hyperbolid, which is a feature that stimulates the proprioceptive function. Thus, this project aims to assess the effects of proprioceptive treatment through the use of hyperbolid on pain intensity, muscle activity and joint mobility in subjects with TMD. A randomized, blind, clinical trial will be conducted. Volunteers aged between 18 and 40 years will be recruited, with a diagnosis of muscle- and joint-related TMD according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC / TMD), being randomly divided in three different groups, the first group constituted by treatment with hyperbolid associated with tongue exercises on the palate, the second group consists of treatment with hyperbolid alone and the third group will not receive any type of intervention (proprioceptive treatment will be offered after the study period). Treatment protocols will be applied for 12 sessions, the volunteers will be evaluated in two stages: before applying the treatment and after the last session. The variables that will be investigated are: pain assessed using visual analog scale and algometry; muscle activity, investigated by electromyography of masticatory muscles; and joint mobility, measured by the use of a caliper. Regarding the analysis of the data will be held intragroup comparisons, considering the pre-treatment and after twelve sessions, and comparisons between groups. To this end it will be applied the Shapiro-Wilk test for checking the normality of data, and the statistical test applied consistent, then parametric or nonparametric. Is assumed a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Temporomandibular Joint Disorders according to the RDC / TMD questionnaire,
* 18 to 40 years

Exclusion Criteria:

* History of neurological disorders
* Submit dental flaws,
* Sull or partial denture,
* Systemic diseases, neuromuscular,
* History of trauma to the face and or ATM
* History of TMJ luxation.
* Being in orthodontic treatment or medication that affects the musculoskeletal system.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 1 Year
  Pain intensity was assessed using the visual analog scale, RDC/TMD Pain Index.

SECONDARY OUTCOMES:
Electromyographic Activity | 1 Year
  Muscle activity was assessed using the EMG signal will be recorded in the dominant upper trapezius muscle in patients with nonspecific neck pain, will be evaluated before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eric Arruda, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

REFERENCES:
- See also: University web site — http://www.uninove.br